CLINICAL TRIAL: NCT03390764
Title: Rein4CeTo1: Incisional Hernia After Colorectal Cancer Surgery - a Randomized Controlled Multicentre Trial Comparing Small Stitch 4:1-technique With Respectively Without a Reinforced Tension-line Suture for Abdominal Closure
Brief Title: Hernia After Colorectal Cancer Surgery
Acronym: Rein4CeTo1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Ulf Petersson, MD, PhD, Ass Prof, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SkaneU
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Incisional Hernia; Wound Dehiscence; Wound Complication; Quality of Life
Keywords: Incisional hernia; 4:1-technique; RTL-suture
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4:1 closure group (Active Comparator): Patients randomized to and receiving the intervention small stitch 4:1 technique for closure of the abdominal wall.
  Interventions: Procedure: 4:1 closure group
- RTL plus 4:1 closure group (Active Comparator): Patients randomized to and receiving the intervention reinforced tension-line suture plus small stitch 4:1 technique for closure of the abdominal wall.
  Interventions: Procedure: RTL plus 4:1 closure group

INTERVENTIONS:
Procedure: 4:1 closure group — In this arm the incisions are closed by the 4:1-technique
  Arms: 4:1 closure group
Procedure: RTL plus 4:1 closure group — In this arm the incisions are closed by a reinforced tension-line suture in addition to the 4:1-technique
  Arms: RTL plus 4:1 closure group

SUMMARY:
Defects in the abdominal wall (incisional hernia) is a frequent negative outcome after surgery. Reinforcing the incision with mesh seem to lower the incidence but in surgery that includes bowel resection a simple alternative, cheaper and less prone to infection than a synthetic mesh, would be of interest. The primary aim of this multicentre randomized controlled trial is to compare the incisional hernia incidence one year after planned colorectal cancer surgery performed through a midline incision which is closed either by a standardized small stitch 4:1 technique (the incision is closed with the use of suture of 4 times the length of the incision) or with the same technique plus a reinforced tension-line suture (a suture is applied in the fibrous tissue parallel to the incision which is then embraced by the 4:1 suture when the incision is closed). A difference in incisional hernia of 15% (20% without and 5% with reinforced tension-line suture) is assumed. Secondary aims are to evaluate incidences of wound dehiscence, other wound complications and incisional hernia after 3 years. Furthermore we aim to evaluate patient satisfaction and quality of life.

DETAILED DESCRIPTION:
The primary aim of this multicentre randomized controlled trial is to compare the incisional hernia incidence one year after planned colorectal cancer surgery performed through a midline incision which is closed either by a standardized small stitch 4:1 technique or with the same technique plus a reinforced tension-line suture. A difference in incisional hernia of 15% (20% without and 5% with reinforced tension-line suture) is assumed and requires inclusion of 76 patients in each group (significance level=5%, power=80%). Patients planned for colorectal surgery due to a cancer are eligible for inclusion. Exclusion criteria are: age below 18, ASA>3, former operation for incisional hernia in the midline, present hernia, perop findings of peritoneal carcinomatosis eligible for peritonealectomy, patient unable to take part in planned follow-up and patient not willing to take part in the study.

Secondary aims are to evaluate incidences of wound dehiscence, other wound complications and incisional hernia after 3 years. Furthermore we aim to evaluate patient satisfaction and quality of life.

Patient base-line characteristics, operative and postop characteristics will be recorded in inclusion- and op-protocols and protocols for clinical follow-up at 1 month, 1 and 3 years. Standard 1 and 3 years CT-scans will be examined for incisional hernia. At 1 and 3 years the patients will be asked to fill out an abdominal wall discomfort enquiry as well as the QoL questionnaire EQ-5D-5L.

The study will be performed at 3 surgical clinics in the Region of Skane in Sweden: Malmö, Kristianstad and Ystad. Inclusion started Oct 2017 and was estimated to be completed after somewhat more than 2 years. The pandemic added 2 years to the inclusion period.The last follow-up will thereby take place after an additional 3 years (2024).

ELIGIBILITY:
Inclusion Criteria:

• Patients ≥ 18 years planned for colorectal cancer surgery through a midline incision

Exclusion Criteria:

* Former incisional hernia surgery in the midline
* Present incisional hernia in the midline
* ASA>3
* Peritoneal carcinomatosis eligible for peritonealectomy/HIPEC
* Patient not able to participate in follow-up
* Patient not willing to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Incisional hernia one year after colorectal cancer surgery comparing a standardized 4:1-technique with and without a reinforced tension-line suture | One year
  Evaluated by clinical investigation and CT-scan

SECONDARY OUTCOMES:
Wound dehiscence and other wound complications | One month or longer
  Early outcome measures investigated during hospitalization and at 1 month follow-up and until wound complication is healed
Incisional hernia after 3 years | 3 years
  Evaluated by clinical investigation and CT-scan
Abdominal wall discomfort at 1- and 3 years follow-up | 1 and 3 years
  Measured by a modified version of the Ventral Hernia Pain Questionnaire
Quality of life after 1- and 3 years | 1 and 3 years
  Measured by the EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Petersson, MD, Ass Prof, Principal Investigator — Department of Surgery, Skane University Hospital, Malmö Sweden
Locations (1):
- Department of surgery, Skane university hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bosanquet DC, Ansell J, Abdelrahman T, Cornish J, Harries R, Stimpson A, Davies L, Glasbey JC, Frewer KA, Frewer NC, Russell D, Russell I, Torkington J. Systematic Review and Meta-Regression of Factors Affecting Midline Incisional Hernia Rates: Analysis of 14,618 Patients. PLoS One. 2015 Sep 21;10(9):e0138745. doi: 10.1371/journal.pone.0138745. eCollection 2015. PMID 26389785
- [Background] Muysoms FE, Dietz UA. Prophylactic meshes in the abdominal wall. Chirurg. 2017 Jan;88(Suppl 1):34-41. doi: 10.1007/s00104-016-0229-7. PMID 27460229
- [Background] Hollinsky C, Sandberg S, Kocijan R. Preliminary results with the reinforced tension line: a new technique for patients with ventral abdominal wall hernias. Am J Surg. 2007 Aug;194(2):234-9. doi: 10.1016/j.amjsurg.2006.09.045. PMID 17618812
- [Background] Agarwal A, Hossain Z, Agarwal A, Das A, Chakraborty S, Mitra N, Gupta M, Ray U. Reinforced tension line suture closure after midline laparotomy in emergency surgery. Trop Doct. 2011 Oct;41(4):193-6. doi: 10.1258/td.2011.110045. Epub 2011 Aug 10. PMID 21831931
- [Background] Millbourn D, Cengiz Y, Israelsson LA. Effect of stitch length on wound complications after closure of midline incisions: a randomized controlled trial. Arch Surg. 2009 Nov;144(11):1056-9. doi: 10.1001/archsurg.2009.189. PMID 19917943
- [Derived] Wenzelberg CL, Rogmark P, Ekberg O, Petersson U. Reinforced tension-line suture after laparotomy: early results of the Rein4CeTo1 randomized clinical trial. Br J Surg. 2024 Sep 3;111(10):znae265. doi: 10.1093/bjs/znae265. PMID 39475416